CLINICAL TRIAL: NCT05030324
Title: A Multicenter, Randomized, Double-blind, Placebo-сontrolled Comparative Study to Evaluate the Safety, Tolerability and Efficacy of XC221 Used at 100 mg Daily and at 200 mg Daily in Patients With Uncomplicated Influenza or Other Acute Viral Upper Respiratory Infections
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of XC221 in Patients With Uncomplicated Influenza or Other Acute Viral Upper Respiratory Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ХС221-02-01-2020
Record Dates: First submitted 2021-08-26; First posted 2021-09-01 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Influenza; Viral Respiratory Infection; Acute Viral Upper Respiratory Infections
Keywords: Influenza; Viral Respiratory Infection; Viral Upper Respiratory Infections; Acute Viral Upper Respiratory Infections; Uncomplicated Influenza
MeSH Terms: conditions — Influenza, Human | interventions — XC221

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into three treatment groups (in a 1:1:1 ratio) receiving: study drug (ХС221) at 100 mg daily or at 200 mg daily, or placebo
Who Masked: Participant, Investigator
Masking Description: Tablets identical in terms of composition, appearance and labeling to XC221 tablets, but without active substance will be used as Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- XC221 100 mg (Experimental): Subjects will receive 1 tablet of XC221, 100 mg tablets orally in the morning (between 7:00 and 11:00) and 1 tablet of placebo in the evening (between 19:00 and 23:00) regardless of food intake for 5 days
  Interventions: Drug: XC221 100 mg
- XC221 200 mg (Experimental): Subjects will receive 1 tablet of XC221, 100 mg tablets orally twice daily, in the morning (between 7:00 and 11:00) and in the evening (between 19:00 and 23:00) regardless of food intake for 5 days
  Interventions: Drug: XC221 200 mg
- Placebo (Placebo Comparator): Subjects will receive 1 tablet of placebo orally twice daily in the morning (between 7:00 and 11:00) and in the evening (between 19:00 and 23:00) regardless of food intake for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XC221 100 mg — Regardless of the group, all study subjects will receive the standard symptomatic therapy for influenza and other viral URIs, taking into account the latest clinical guidelines (the necessity of symptomatic therapy will be decided by the Investigator).
  Arms: XC221 100 mg
Drug: XC221 200 mg — Regardless of the group, all study subjects will receive the standard symptomatic therapy for influenza and other viral URIs, taking into account the latest clinical guidelines (the necessity of symptomatic therapy will be decided by the Investigator).
  Arms: XC221 200 mg
Drug: Placebo — Regardless of the group, all study subjects will receive the standard symptomatic therapy for influenza and other viral URIs, taking into account the latest clinical guidelines (the necessity of symptomatic therapy will be decided by the Investigator).
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, placebo controlled comparative study to evaluate the safety, tolerability and efficacy of XC221 used at 100 mg daily and at 200 mg daily in patients with uncomplicated influenza or other acute viral upper respiratory infections (URIs) for 5 days of treatment.

The primary objective of the study is to evaluate the efficacy of ХС221 at 100 mg and at 200 mg in comparison with placebo regarding its effect on the severity and duration of influenza symptoms and symptoms of other viral URIs (fever and other major signs and symptoms).

The secondary objective of the study is to evaluate the safety of ХС221 at 100 mg and at 200 mg in comparison with placebo in the treatment of influenza ad other viral URIs.

DETAILED DESCRIPTION:
Russian centers will participate in this study. This is a double-blind, placebo-control study, and therefore, in order to maintain the study design, subjects will be administered with placebo or the study drug depending on the treatment group they have been randomized into.

The screening visit and all other visits of the study will be on an outpatient basis (including home visits). The study will consist of three periods: screening, randomization and initiation of treatment ( Day 1); treatment period (Day 1-5) and follow-up period (Day 6-20± 1 after completion of treatment with XC221 / Placebo). The duration of participation in the study for each patient will be no more than 21 days.

255 eligible patients will be randomized into three treatment groups (in a 1:1:1 ratio) and receive: study drug (ХС221) at 100 mg daily or at 200 mg daily, or placebo. Regardless other group, all study subjects should receive the standard symptomatic therapy for influenza and other viral URIs, taking into account the latest clinical guidelines (the necessity of symptomatic therapy will be decided by the Investigator).

Group 1: subjects will receive 1 tablet of XC221, 100 mg tablets orally in the morning (between 7:00 and 11:00) and 1 tablet of placebo in the evening (between 19:00 and 23:00) regardless of food intake for 5 days.

Group 2: subjects will receive 1 tablet of XC221, 100 mg tablets orally twice daily in the morning (between 7:00 and 11:00) and in the evening (between 19:00 and 23:00) regardless of food intake for 5 days.

Group 3: subjects will receive 1 tablet of placebo orally twice daily, in the morning (between 7:00 and 11:00) and in the evening (between 19:00 and 23:00) regardless of food intake for 5 days.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 65 years (inclusive);
2. Signed Informed Consent Form;
3. Clinical symptoms of mild to moderate influenza and other viral URIs:

   * an increased axillary temperature of ≥38.0°С ≤39.5°С during the current illness without the use of antipyretics in the last 8 hours at the time of screening;
   * at least one of the respiratory signs and symptoms of influenza or other viral URIs (cough, runny nose/nasal congestion, sore throat) scored at least 2 points on a 4-point scale;
   * at least one of the systemic signs and symptoms of influenza or other viral URIs (headaches, muscle aches, chills/sweats, fatigue) scored at least 2 points on a 4-point scale.
4. Absence of indications for hospitalization at the time of enrollment;
5. Duration of illness from symptom manifestation to the first drug dose/placebo no more than 48 h;
6. Negative pregnancy test for women of childbearing potential;
7. A consent to use adequate birth control methods throughout the treatment and for 30 days thereafter;
8. Patients who are able to understand and comply with treatment and procedures during the study.

Exclusion Criteria:

1. Pregnant and lactating women;
2. Known or suspected hypersensitivity to the active substance or to excipients of the drug XC221 or placebo;
3. An established or currently suspected diagnosis (based on the assessment of the patient's health and epidemiological medical history) of COVID-19;
4. Oxygen saturation (SpO2) ≤ 95%, respiration rate (RR) ≥ 22/min.
5. Complications of influenza or other viral URIs;
6. Participation in another clinical trial within 90 days prior to screening;
7. Known (based on the medical history) or suspected abuse of alcohol or psychotropic drugs;
8. Patients with psychotic diseases, including in the medical history;
9. Moderate viral URI (fever ≥ 38.5°С) accompanied by exacerbation of concomitant conditions;
10. Clinically suspected pneumonia or other bacterial infections (including sinusitis, otitis media, urinary tract infection, meningitis, sepsis, etc.) requiring antibacterial therapy;
11. Taking antibiotics, antivirals, or immunomodulatory drugs within < 48 h prior to treatment initiation and/or planning to use these types of drugs (except for the investigational products) during the study;
12. Use of systemic, inhaled or nasal corticosteroids within 30 days prior to treatment initiation and/or planning to use corticosteroids (except for topical dermatological agents) during the study;
13. The inability to cancel during the study period other drugs that can affect the result of this study, for example, antiviral drugs, or drugs that are incompatible with the study's therapy;
14. Any diseases of cardiac, renal, hepatic, gastrointestinal, endocrine and nervous system, severe decompensated chronic (including chronic renal and liver diseases) or acute diseases, or any other conditions/diseases which would make participation in the study unsafe (in the investigator's opinion);
15. Patients receiving any vaccines within 90 days prior to enrollment;
16. Diabetes mellitus, grade 2-3 obesity;
17. Patients who underwent surgery within 30 days prior to the screening and patients who are scheduled to undergo surgery during the study period, including diagnostic procedures or hospital stay;
18. Patients with oncological diseases, HIV infection, or tuberculosis, including a medical history;
19. Meningeal syndrome;
20. Disorders of consciousness (in the form of stupor, sopor, delusion, delirium, etc.);
21. Symptoms of pneumonia and possible acute respiratory distress syndrome (ARDS): cough with bloody frothy sputum, shortening of pulmonary sound with percussion, a large number of different-sized wet wheezing and profuse crepitus on auscultation, a sharp decrease in blood pressure (BP), deafness of heart sounds and arrhythmia;
22. Positive rapid test result for SARS-CoV-2;
23. Lactase deficiency, lactose intolerance, glucose-galactose malabsorption.
24. Other reasons which would prevent the patient from participating in the study and make an unreasonable risk (in the investigator's opinion).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Time (in hours) from the first dose of the drug to the resolution of all of the following symptoms/events. | Day 1 - Day 10
  • fever (the day of fever resolution is the first day on which stable normal body temperature is achieved (<37.0°C without the use of antipyretics));
  All achieved symptoms/events scores maintained for at least 24 h at 0-1 point:
  * nasal congestion/runny nose;
  * sore throat;
  * cough;
  * muscle aches;
  * headaches;
  * fatigue;
  * chills/sweats.
  Patients will assess and record the severity of all symptoms on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.

SECONDARY OUTCOMES:
Time to decrease in 24-hour body temperature to ≤ 37.0°C without using antipyretics (number of hours from the first dose of the study treatment to a decrease in 24-hour body temperature to ≤ 37.0°C). | Day 1 - Day 10
  Patients will assess and record body temperature in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents.
Time to nasal congestion/runny nose resolution (number of hours from the first dose of the drug to runny nose/congestion resolution, i.e. the time when the subject rates the 24-hour severity of this symptom at 0-1 point) | Day 1 - Day 10
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom
Patient rate with reported nasal congestion/runny nose resolution by day 4 and day 6 from treatment initiation (i.e. patient rate who assessed the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 6
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Time to sore throat resolution (number of hours from the first dose of the drug to sore throat resolution, i.e. the time when the subject rates the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 10
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Patient rate with reported sore throat resolution by day 4 and day 6 from treatment initiation (i.e. patient rate who assessed the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 6
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Time to cough resolution (number of hours from the first dose of the drug to cough resolution, i.e. the time when the subject rates the 24-hour severity of this symptom at 0-1 point. | Day 1 - Day 10
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Patient rate with reported cough resolution by day 4 and day 6 from treatment initiation (i.e. patient rate who assessed the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 6
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Time to muscle ache resolution (number of hours from the first dose of the drug to the resolution of muscle aches, i.e. the time when the subject rates the 24-hour severity of this symptom at 0-1 point | Day 1 - Day 10
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Patient rate with reported muscle ache resolution by day 4 and day 6 from treatment initiation (i.e. patient rate who assessed the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 6
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Time to headache resolution (number of hours from the first dose of the drug to headache resolution, i.e. the time when the subject rates the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 10
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Patient rate with reported headache resolution by day 4 and day 6 from treatment initiation (i.e. patient rate who assessed the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 6
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Time to fatigue resolution (number of hours from the first dose of the drug to fatigue resolution, i.e. the time when the subject rates the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 10
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Patient rate with reported fatigue resolution by day 4 and day 6 from treatment initiation (i.e. patient rate who assessed the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 6
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Time to chills/sweats resolution (number of hours from the first dose of the drug to the resolution of chills/sweats, i.e. the time when the subject rates the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 10
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Patient rate with reported chills/sweats resolution by day 4 and day 6 from treatment initiation (i.e. patient rate who assessed the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 6
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Frequency complications of influenza or other viral URIs (sinusitis, otitis, bronchitis, pneumonia). | Day 1 - Day 10
Time till elimination viruses based on qualitative PCR test (i.e. time to the first negative PCR test). | Day 1 - Day 10
The need for paracetamol or ibuprofen: daily dose on days 1-10. | Day 1 - Day 10

CONTACTS AND LOCATIONS:
Locations (9):
- Russia (9):
  - State autonomous health care institution "Engels City Clinical Hospital No. 1", Engel's
  - Limited Liability Company "Health Energy", Saint Petersburg
  - Limited Liability Company "MEDICAL CLINIC", Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Polyclinic No. 117", Saint Petersburg
  - Saint Petersburg State Budgetary Healthcare Institution "City polyclinic No. 112", Saint Petersburg
  - Limited Liability Company "Research Center Eco-Security", Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Polyclinic No. 4", Saint Petersburg
  - Limited Liability Company "Meili", Saint Petersburg
  - State budgetary institution of health care of the Yaroslavl region "Clinical Hospital No. 2", Yaroslavl

IPD SHARING:
Plan to Share IPD: No